CLINICAL TRIAL: NCT06063577
Title: A Randomized Controlled Trial Evaluating the Use of Stratafix Symmetric™ to Prevent Incisional Hernia in Gastrointestinal and Abdominal Surgery
Brief Title: Use of Stratafix Symmetric™ to Prevent Incisional Hernia in Gastrointestinal and Abdominal Surgery
Acronym: STRATA-G
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Michigan Cancer Center (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Gitonga Munene, Principal Investigator, West Michigan Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001-2023
Record Dates: First submitted 2023-09-02; First posted 2023-10-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: C.Surgical Procedure; Disruption of Wound, Suture

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded after the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Stratafix Group (Active Comparator): Stratafix
  Interventions: Device: Stratafix suture
- Control Group (Placebo Comparator): Standard of care
  Interventions: Device: Standard of care suture

INTERVENTIONS:
Device: Stratafix suture — Stratafix symmetric suture
  Arms: Stratafix Group
Device: Standard of care suture — Standard of care suture
  Arms: Control Group

SUMMARY:
Comparing the use of Stratafix Symmetric™ sutures to standard laparotomy closure sutures.

DETAILED DESCRIPTION:
Determine whether the use of Stratafix Symmetric™ sutures reduces the development of Ventral Incisional Hernia (VIH) in patients undergoing complex GI surgery compared to standard laparotomy closure. Determine the safety of Stratafix Symmetric™ sutures compared to standard laparotomy closure sutures and the impact on quality of life and level of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a male or female 18 years of age or older.
2. Participant is a current patient at West Michigan Cancer Center.
3. Participant is undergoing liver, pancreas or biliary or gastrointestinal surgery of a combination of the above, or other major oncological surgery.
4. Participant is willing and able to provide written informed consent before surgery.

Exclusion Criteria:

1. Participant has hemodynamic instability at the conclusion of the surgery. (These subjects will be deemed disqualified).
2. Participant has history of previous VIH.
3. Participant has a mental condition rendering the subject incapable of understanding the nature, scope and consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop ventral incisional hernia | From enrollment to end of study participation at 12 months
  Infection, seroma, surgical site infection, evisceration, mesh rejection, systemic complications

SECONDARY OUTCOMES:
Safety of stratafix sutures compared to standard of care wound closure | From enrollment to end of study participation at 12 months
  Assessing adverse events related to the suture
Change in quality of life | "Month 1," "Month 3," "Month 6," "Month 12"
  Carolinas Comfort Scale (CCS) questionnaire (a validated, disease-specific, quality of life (QOL) questionnaire developed for patients undergoing hernia repair)
Change in quality of life | "Day 1," "Month 1," "Month 3," "Month 6," "Month 12"
  Functional Assessment of Cancer Therapy-G (FACT-G) questionnaire (a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being.)
Post operative pain | From enrollment to end of study participation at 12 months
  Visual analog score

CONTACTS AND LOCATIONS:
Overall Officials: Gitonga Munene, Principal Investigator — West Michigan Cancer Center
Locations (1):
- West Michigan Cancer Center, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No